CLINICAL TRIAL: NCT04219475
Title: Predicting Response Patterns to Treatment in Glioblastoma (GBM) Oncology Patients Based on Host Response Evaluation During Anti-cancer Treatments
Brief Title: Predicting Response Patterns to Treatment in Glioblastoma (GBM) Patients
Acronym: PROPHETIC
Status: Suspended | Type: Observational
Why Stopped: Priority changes of the company
Sponsor: OncoHost Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: OH-GBMHR
Record Dates: First submitted 2019-12-31; First posted 2020-01-07 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GBM patients: Newly diagnosed patients above 18 years of age with GBM receiving standard of care, i.e., maximal surgical resection possible followed by radiation therapy (RT) plus temozolomide (TMZ) therapy and maintenance TMZ.

SUMMARY:
PROPHETIC GBM - Predicting response patterns to treatment in Glioblastoma (GBM) oncology patients based on host response evaluation during anti-cancer treatments

DETAILED DESCRIPTION:
The goal of this research study is identify new host response proteins, pathways and mechanisms that are associated with responsiveness to GBM treatment modalities.

This will serve as a tool for physicians when making treatment decisions. The investigators also aim to identify the metabolic pathways that could lead to better therapeutic options. The patients will be given their treatment according to the institute's standard of care. The patients will provide up to 5 blood samples and clinical data will be collected from their medical records.

The data obtained from the blood samples and the medical records of the patients will be used to search for potential mechanisms that are involved in response to treatment, and to identify potential targets to increase the response, and hence, increase treatment effectiveness or suggest potential new treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study-specific procedures.
2. Male or female aged at least 18 years.
3. KPS not less than 50.
4. Normal hematologic, renal and liver function:

   1. Absolute neutrophil count above 1500/mm3, platelets above 100,000/mm3, hemoglobin above 9 g/dL;
   2. Creatinine concentration not more than 1.4 mg/dL, or creatinine clearance above 40 mL/min;
   3. Total bilirubin below 1.5 mg/dL, ALT+ AST levels not more than 3 times above the upper normal limit.
5. Patients planned to receive standard of care TMZ+RT treatment; TTF therapy during RT is permitted.

Exclusion Criteria:

1. Any concurrent and/or other active malignancy that has required systemic treatment within 2 years of surgery. Except for basal cell carcinomas and squamous cell carcinomas that have been completely excised and considered cured at least 12 months prior to screening, and carcinoma in situ of the cervix that have been completely excised and cured at least 5 years prior to screening.
2. Participation in another clinical trial which includes an investigational drug.
3. Generalized impairment or mental incompetence that would render the patient unable to understand his/her participation in the study.
4. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients recruited for the study except for
  1. Patients who discontinued the TMZ during the first 2 weeks of treatment, unless the drug was stopped due to tumor progression.
  2. Patients who didn't receive at least 46 Gy in the 6 weeks regimen or 30 Gy in the 3 weeks regimen, unless the treatment was stopped due to grade 3 and higher toxicity.
  3. Patients who chose to discontinue the treatment for reasons other than disease progression or serious side effects unless the treatment was stopped due to grade 3 and highertoxicity.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Response to treatment | One month after completion of TMZ + RT
  complete remission (CR); partial remission (PR), stable disease (SD), progressive disease (PD), suspected pseudo-progression, as defined by RANO
Response to treatment | 3 months after treatment completion in the first year
  CR, PR, SD, PD, suspected pseudo-progression, as defined by RANO
Response to treatment | 6 months after treatment completion in the first year
  CR, PR, SD, PD, suspected pseudo-progression, as defined by RANO
Response to treatment | 9 months after treatment completion in the first year
  CR, PR, SD, PD, suspected pseudo-progression, as defined by RANO
Response to treatment | 12 months after treatment completion in the first year
  CR, PR, SD, PD, suspected pseudo-progression, as defined by RANO
Response to treatment | 18 months after treatment completion in the first year
  CR, PR, SD, PD, suspected pseudo-progression, as defined by RANO
Response to treatment | 24 months after treatment completion in the first year
  CR, PR, SD, PD, suspected pseudo-progression, as defined by RANO
Response to treatment | 30 months after treatment completion in the first year
  CR, PR, SD, PD, suspected pseudo-progression, as defined by RANO
Response to treatment | 36 months after treatment completion in the first year
  CR, PR, SD, PD, suspected pseudo-progression, as defined by RANO
Blood levels of proteins | Pre-chemoradiation therapy - 7 days or less before the first administration
  Blood levels of proteins representing the Host response at baseline
Blood levels of proteins | After the first chemoradiation administration - at least 24 h after the first temozolomide (TMZ) dose, and between 24-48 h after the first radiation therapy (RT) dose
  Changes in Blood levels of proteins representing the Host response compared to baseline
Blood levels of proteins | 21+/-2 days after the first TMZ dose
  Changes in Blood levels of proteins representing the Host response compared to baseline
Blood levels of proteins | At first detection of progressive disease (PD) based on MRI evaluation during follow-up assessed up to 36 months
  Changes in Blood levels of proteins representing the Host response compared to baseline
Blood levels of proteins | If the previous detection of progression turned out to be pseudo-progression, then an additional blood sample should be drawn at time of progression, assessed up to 36 months
  Changes in Blood levels of proteins representing the Host response compared to baseline

SECONDARY OUTCOMES:
OS | Until death or 3 years
  Overall survival
PFS | up to 3 years
  Progression free survival

CONTACTS AND LOCATIONS:
Overall Officials: Dror Limon, MD, Principal Investigator — Sourasky Medical Center
Locations (4):
- Israel (4):
  - Rambam medical center, Haifa
  - Rabin medical center, Petah Tikva
  - Sourasky medical center, Tel Aviv
  - Sheba medical center, Tel Litwinsky

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shaked Y. Balancing efficacy of and host immune responses to cancer therapy: the yin and yang effects. Nat Rev Clin Oncol. 2016 Oct;13(10):611-26. doi: 10.1038/nrclinonc.2016.57. Epub 2016 Apr 26. PMID 27118493
- [Background] Shaked Y, Kerbel RS. Antiangiogenic strategies on defense: on the possibility of blocking rebounds by the tumor vasculature after chemotherapy. Cancer Res. 2007 Aug 1;67(15):7055-8. doi: 10.1158/0008-5472.CAN-07-0905. PMID 17671170
- [Background] Shaked Y, Bocci G, Munoz R, Man S, Ebos JM, Hicklin DJ, Bertolini F, D'Amato R, Kerbel RS. Cellular and molecular surrogate markers to monitor targeted and non-targeted antiangiogenic drug activity and determine optimal biologic dose. Curr Cancer Drug Targets. 2005 Nov;5(7):551-9. doi: 10.2174/156800905774574020. PMID 16305351